CLINICAL TRIAL: NCT01502397
Title: Risk of Hepatitis B Reactivation in Patients With Prior HBV Exposure Undergoing Rituximab-containing Chemotherapy: A Prospective Study
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: HKCTR-1431; HKCTR-1431 (Registry Identifier: HKU CTC)
Record Dates: First submitted 2011-12-28; First posted 2011-12-30 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Exposure to Hepatitis B Virus
Keywords: hepatitis B; anti-HBc; HBsAg; rituximab; occult HBV
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma for hepatitis B virus genotypic, virologic and serologic testing
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HBsAg-negative, anti-HBc-positive: HBsAg-negative, anti-HBc-positive subjects undergoing rituximab-containing chemotherapy

SUMMARY:
The purpose of this study is to determine whether preemptive nucleoside analogue therapy or regular virologic monitoring is the preferred method in management patients with prior exposure to hepatitis B vius (HBV) and undergoing rituximab-containing chemotherapy.

DETAILED DESCRIPTION:
Occult hepatitis B virus (HBV) reactivation has been documented in patients undergoing rituximab-containing chemotherapy who are hepatitis B surface antigen (HBsAg)-negative but with serologic evidence of prior exposure to HBV. However detailed prospective studies documenting the incidence of reactivation and the virologic and serologic kinetics of reactivation are lacking. The investigators prospective study proposes to follow-up 70 such patients with all serologic and virologic parameters monitored every 4 weeks. Patients with detectable HBV DNA will be started on nucleoside analogue therapy. The optimal method and duration of monitoring will also be determined from our study.

ELIGIBILITY:
Inclusion Criteria:

* Documented HBsAg-negative with or without antibody to hepatitis B surface antigen (anti-HBs)
* Documented anti-HBc (total)-positive

Exclusion Criteria:

* Concomitant liver diseases including chronic hepatitis C and D infection, Wilson's disease, autoimmune hepatitis, primary biliary cirrhosis and primary sclerosing cholangitis.
* Significant alcohol intake (>30 grams per day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with B-cell lymphomas or chronic lymphocytic leukaemia referred to Queen Mary Hospital for rituximab-containing chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
HBV reactivation (defined as detectable HBV DNA > 20 IU/mL) | 2 years
  From date of rituximab commencement up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Man-Fung Yuen, FRCP, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Medicine, The University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong